CLINICAL TRIAL: NCT01782937
Title: A Long-Term Study of KHK4827 in Subjects With Pustular Psoriasis (Generalized) and Psoriatic Erythroderma
Brief Title: An Open-label, Non-controlled Study of KHK4827 in Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4827-004
Record Dates: First submitted 2013-01-27; First posted 2013-02-04 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KHK4827 (Experimental)
  Interventions: Drug: KHK4827

INTERVENTIONS:
Drug: KHK4827 — 140 mg (dosage may be increased to 210 mg in case of insufficient efficacy)

SUMMARY:
This study is an open-label, non-controlled study to evaluate the efficacy and safety of KHK4827 in subjects with pustular psoriasis (generalized) and psoriatic erythroderma. Pharmacokinetics of KHK4827 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed voluntarily the written informed consent form to participate in this study.
* Subject has been diagnosed as pustular psoriasis or psoriatic erythroderma.
* Subject has received at least one previous phototherapy or systemic psoriasis therapy or has been a candidate to receive phototherapy or systemic psoriasis therapy in the opinion of the investigator.

Exclusion Criteria:

* Subject with psoriatic erythroderma has involved Body surface area (BSA) of lesion < 80% at baseline.
* Subject diagnosed with guttate psoriasis, medication-induced or medication-exacerbated psoriasis.
* Evidence of skin conditions at the time of the screening visit (eg, eczema) that would interfere with evaluations of the effect of KHK4827 on psoriasis.
* Subject has any active Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher infection
* Subject has a significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol.
* Subject has used Ultra Violet B (UVB) therapy within 14 days of the first dose or Ultra Violet A (UVA) (with or without psoralen) within 28 days of the first dose.
* Subject has used etanercept, adalimumab, infliximab or ustekinumab within 1 week, 2 weeks, 8 weeks or 12 weeks of the first dose, respectively.
* Subject has stopped ustekinumab or other anti-Interleukin (IL)-23 biologics therapy due to lack of efficacy
* Subject has used live vaccine within 3 months of the first dose
* Subject has previously used an anti-IL-17 biologic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) | 52 weeks
  CGI is a 4-point scale that requires the investigators/subinvestigators to assess how much the subject's illness has improved or worsened relative to a baseline state. Scores on the scale are rated as: 1, remission; 2, improved; 3, no change; 4, worsened

SECONDARY OUTCOMES:
Percent improvement from baseline in Psoriasis Area and Severity Index (PASI) | 52 weeks
American College of Rheumatology (ACR) 20 (only in subjects with psoriasis arthritis) | 52 weeks
Pustular symptom score (only in subjects with pustular psoriasis) | 52 weeks
Static physician's global assessment (sPGA) of "clear or almost clear (0 or 1)" at Week 12 (only in subjects with psoriatic erythroderma) | 52 weeks
sPGA of "clear (0)" at Week 12 (only in subjects with psoriatic erythroderma) | 52 weeks
Body surface area involvement (BSA) of lesion at Week 12 (only in subjects with psoriatic erythroderma) | 52 weeks
Incidence and types of adverse events and adverse reactions | 52 weeks
Laboratory values and vital signs | 52 weeks
Profiles of pharmacokinetics | 52 weeks
  Concentration of KHK4827 in serum
Development of anti-KHK4827 antibody | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Chiyoda-ku, Tokyo, Japan